CLINICAL TRIAL: NCT05304364
Title: Open-Label Study in Healthy Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics of Switching From Oral Naltrexone HCL to DLP-160 (Naltrexone Implant) to Intramuscular Vivitrol®
Brief Title: Safety, Tolerability, and Pharmacokinetics of Naltrexone Implant (DLP-160)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Delpor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DLP-160-01
Record Dates: First submitted 2022-03-07; First posted 2022-03-31 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Opiod Use Disorder
Keywords: Naltrexone; Addiction; Mental Health; Implant
MeSH Terms: conditions — Behavior, Addictive; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DLP-160 alpha-10 (Experimental): One time single Naltrexone Implant for a duration of 123 days
  Interventions: Combination Product: Combination Product: Naltrexone

INTERVENTIONS:
Combination Product: Combination Product: Naltrexone — Naltrexone Implant
  Other Names: DLP-160

SUMMARY:
This is an Open-Label Study in Healthy Volunteers to Evaluate the Safety, Tolerability, and Pharmacokinetics of Switching from Oral Naltrexone HCL to DLP-160 (Naltrexone implant) to Intramuscular Vivitrol®

DETAILED DESCRIPTION:
This study is first-in-man clinical study of DLP-160, a Naltrexone implant product. The study is an open-label, single sequence design aimed at assessing the safety and tolerability of DLP-160 and evaluating its utility in achieving a PK profile that is comparable to the marketed oral and injectable forms of Naltrexone.

Initially, a group of 2 healthy volunteers will receive the Naltrexone HCL followed by DLP-160 implant as a sentinel group. The safety and tolerability of the DLP-160 implant will be assessed in the sentinel group for at least 28 days prior to any other volunteers being implanted with DLP-160 in the study. Only if the safety and tolerability data, obtained from the sentinel group, are considered acceptable by the Investigator, will the remainder of healthy volunteers commence treatment in the study.

Healthy volunteers will be enrolled and implanted with DLP-160 involving treatment of each study participant consisting of 3 sequential treatment periods with a washout period between treatments.

1. Naltrexone HCL treatment (oral; 50 mg/day) (Day -6 to Day -2);
2. Washout (Day -1);
3. DLP-160 implant treatment (up to 123 days);
4. DLP-160 removal and washout (1 day);
5. Vivitrol® treatment (single intramuscular injection with a 30 day follow up);
6. Follow up to completion of study participation (7 days).

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 50 years of age (inclusive) at the time of screening.
3. Body Mass Index (BMI) greater than or equal to 18.0 and lesser than or equal to 30.0 kg/m2, with a body weight (to 1 decimal place) greater than or equal to 50 kg.
4. Medically healthy without clinically significant abnormalities (in the opinion of the Investigator) at the screening visit and prior to administration of the first study dose on study Day -6, including:

   1. Physical examination without any clinically significant findings.
   2. Systolic blood pressure in the range of 90 to 160 mmHg (inclusive) and diastolic blood pressure in the range of 50 to 95 mmHg (inclusive) after 5 minutes in supine (or semi-supine) position.
   3. Heart rate (HR) in the range of 45 to 100 bpm (inclusive) after 5 minutes rest in a supine (or semi-supine) position.
   4. Body temperature (tympanic or oral) in the range 35.5°C to 37.7°C (inclusive).
   5. No clinically significant findings in serum chemistry, haematology, coagulation, and urinalysis tests.
   6. Triplicate 12-lead ECG (taken after the volunteer has been supine (or semi-supine) for at least 5 minutes) with a QT interval corrected using the Fridericia method (QTcF) lesser than or equal to 450 msec for males and lesser than or equal to 470 msec for females and no clinically significant abnormalities.

   Note: Minor abnormalities or deviations outside the normal ranges for any of the clinical testing (laboratory tests, ECG, vital signs) may be repeated at the discretion of the Investigator. Such abnormalities or deviations are acceptable for participation in the study if judged to be not clinically significant by the Investigator. Platelet count and coagulation measures must be within normal limits.
5. Female volunteers must:

   1. Be of nonchildbearing potential i.e., be surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or be postmenopausal, where menopause is defined as 12 months of amenorrhea in the absence of other biological causes (females under the age of 55 years must have a documented serum follicle stimulating hormone (FSH) level greater than 40mIU/mL to confirm menopause).
   2. If of childbearing potential (defined as any female who has experienced menarche and who has not undergone surgical sterilisation and is not postmenopausal), the participant:

      * Must have a negative serum test at the screening visit and a negative urine pregnancy test within 24 hours prior to the start of study drug.
      * Must not be breastfeeding, lactating or planning pregnancy during the study period.
      * Must agree not to attempt to become pregnant.
      * If not exclusively in same-sex relationships, must agree to use adequate contraception (which is defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner); after signing consent, during the study, and at least 35 days after the last dose of study drug;
      * Must agree to not donate ova for at least 35 days after the last dose of study drug.
6. Male participants, if not surgically sterilised, must agree to:

   1. Not donate sperm after signing consent, during the study, and at least 95 days after the last dose of study drug.
   2. If engaging in sexual intercourse with a female partner who could become pregnant, use a condom in addition to having the female partner use a highly effective contraceptive method.
   3. Have suitable venous access for blood sampling.
7. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the past 3 months determined by the PI to be clinically significant (participants with resolved childhood asthma may be included in the study).
2. Current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic or antiviral medications.
3. Liver function test results elevated more than 1.5-fold above the upper limit of normal (ULN) for gamma glutamyl transferase (GGT), bilirubin (total, conjugated and unconjugated), alkaline phosphatase (ALP), aspartate aminotransferase (AST) or alanine aminotransferase (ALT). Volunteers with ALP and/or ALT/AST above the limits specified may be included, at the discretion of the Investigator, if the levels are unaccompanied by clinical signs and are determined to be normal variants.
4. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at the screening visit.
5. Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs (prior gall bladder and/or appendix removal is not exclusionary if deemed appropriate by the Investigator).
6. Estimated creatinine clearance (CrCl) less than 80 mL/min using the Cockcroft-Gault formula or serum creatinine more than 1.5-fold above the ULN.
7. Presence of clinically significant skin disorders (such as, but not limited to, skin cancer, psoriasis, eczema, or atopic dermatitis), evidence of recent sunburn, scar tissue, tattoo, open sore, body piercing or branding at the intended placement site that would interfere with the placement procedure or interfere with implant site assessments as determined by the Investigator.
8. History of abnormal scar formation or family history of keloid formation.
9. Known hypersensitivity to titanium, implant materials or the procedure of implant placement.
10. Previously defined hypersensitivity to Naltrexone.
11. Known hypersensitivity or allergy to lidocaine or any local anaesthetic agent of the amide type (local anaesthetic used during placement and removal procedures).
12. History of substance abuse, in the opinion of the Investigator.
13. History of alcohol abuse (defined as more than an average of 14 standard drinks per week or regular consumption of more than 4 standard drinks on any one day; where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc./Vol], 100 mL wine [12% Alc./Vol], 30 mL spirit [40% Alc./Vol]).
14. Positive drugs of abuse or alcohol breath test results at the screening visit or prior to the first study drug administration on Day -6 and at check-in on Day -2.
15. Use of any prescription or over-the-counter medication (including herbal products, and hormone supplements) within 10 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration - exceptions include contraceptives for females, occasional use of paracetamol (doses of 500 mg up to every 6 hours or 2 g per day maximum for no more than 3 consecutive days), ibuprofen (doses of 400 mg up to every 6 hours or 1.2 g per day maximum for no more than 3 consecutive days), topical ointments, and vitamins or dietary supplements.
16. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the trial.
17. For women of childbearing potential, a positive serum pregnancy test at the screening visit or a positive urine pregnancy test (with confirmatory serum pregnancy test) prior to the first study drug administration on Day -6 and at check-in on Day -2.
18. Females who are breastfeeding or planning to breast feed at any time during the study.
19. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to first study drug administration, or receipt of a blood transfusion within 1 year of first study drug administration.
20. Intolerance of direct venepuncture.
21. Treatment with an investigational drug (or device) in another clinical trial within 30 days or 5 half-lives of the other investigational drug (whichever is longer) prior to the first administration of study drug in this trial.
22. Anticipated surgical procedure or current painful condition that is likely to require opioid analgesia during the trial.
23. Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-11-19 (Actual)

PRIMARY OUTCOMES:
DLP-160 Adverse Events | Day 1 to Day 120
  Determine the number and percent of patients experiencing a treatment-emergent adverse event
DLP-160 Local Tolerance | Day 1 to Day 120
  Evaluate the incidence of local site reactions
Tolerability of DLP-160 Implantation and Removal Procedures | Day 1 to Day 120
  Assess the incidence of local site reactions and/or Adverse Events (AEs) reported during the implantation and removal procedure

SECONDARY OUTCOMES:
Oral Pharmacokinetic (PK) Profile | 24 hours
  Measure the plasma concentration of Naltrexone, 6-β-naltrexol and active moiety (Naltrexone + 6-β-naltrexol) following:
  • Repeated oral administrations Naltrexone HCL
Implant Pharmacokinetic (PK) Profile | 4 months
  Measure the plasma concentration of Naltrexone, 6-β-naltrexol and active moiety (Naltrexone + 6-β-naltrexol) following:
  • Following treatment switch from oral Naltrexone HCL to subcutaneous placement of one DLP-160 implant
IM Naltrexone PK Profile | 1 month
  Measure the plasma concentration of Naltrexone, 6-β-naltrexol and active moiety (Naltrexone + 6-β-naltrexol) following:
  • Following treatment switch from one DLP-160 implant to a single IM dose of Vivitrol®.
Evaluate the Drug Output of the DLP-160 Implant | 4 months
  Evaluate the amount of Naltrexone drug substance remaining in the DLP-160 implant drug reservoir following its removal and estimating daily drug output of the DLP-160 implant.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Choo, MD, Principal Investigator — CMAX
Locations (1):
- CMAX, Adelaide, South Australia, Australia